CLINICAL TRIAL: NCT01699542
Title: A Multi-Center, Prospective, Randomized (RCT) Study Comparing WallFlex® Esophageal Fully Covered (FC) Metal Stent to Bougie Dilation for the Treatment of Refractory Anastomotic Esophageal Strictures
Brief Title: WallFlex Esophageal Fully Covered (FC) Benign Anastomotic Stricture
Acronym: E7025
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90913904
Record Dates: First submitted 2012-10-02; First posted 2012-10-03 (Estimated); Results first posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-04

CONDITIONS: Refractory Anastomotic Esophageal Strictures
Keywords: Refractory Anastomotic esophageal strictures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metal Stent (Active Comparator): The WallFlex Biliary Fully Covered Esophageal Stent System is being evaluated for treatment of refractory anastomotic esophageal strictures.
  Interventions: Device: WallFlex Esophageal RX Fully Covered Stent
- Bougie Dilation (Active Comparator): Esophageal Bougie Dilator commercially available devices used per Investigator preference are being evaluated for treatment of refractory anastomotic esophageal strictures.
  Interventions: Device: Esophageal Bougie Dilator Per Investigator preference

INTERVENTIONS:
Device: WallFlex Esophageal RX Fully Covered Stent — Temporary placement of the WallFlex Esophageal RX Fully Covered Stent for treatment of refractory anastomotic esophageal strictures. The stent will be removed after 8 weeks (plus or minus 7 days) indwell
  Arms: Metal Stent
Device: Esophageal Bougie Dilator Per Investigator preference — Commercially available Esophageal Bougie Dilator Per Investigator preference
  Arms: Bougie Dilation

SUMMARY:
The purpose of this of this study is to compare the safety and effectiveness of temporary indwell of the WallFlex Esophageal FC Metal Stent to Bougie Dilation for the treatment of refractory anastomotic esophageal strictures

ELIGIBILITY:
Inclusion Criteria:Esophageal anastomotic stricture post esophagectomy (esophagogastric strictures).

* Esophagectomy performed at the same institution where patient enrollment and follow-up is planned.
* Two dilations to at least 16 mm in diameter since esophagectomy.
* 1st dilation no more than 6 months post esophagectomy and 2nd dilation within 6 months of 1st dilation to 16mm.
* Dysphagia score of 2 (ability to swallow semi-solid foods), 3 (ability to swallow liquids only) or 4 (unable to swallow liquids) at baseline.
* Unable to pass a standard endoscope (approx. 9.8 mm diameter).
* Age 18 years or older.
* Willing and able to comply with the study procedures and provide

Exclusion Criteria:Stricture within 2 cm of the upper esophageal sphincter.

* Dysphagia related to motility disorder.
* Non-anastomotic esophageal strictures.
* Esophagocolonic strictures.
* Planned adjuvant radiation therapy post esophagectomy.
* Prior esophageal stent placements post esophagectomy.
* Active erosive esophagitis.
* Sensitivity to any components of the stent or delivery system.
* Concurrent medical condition that would affect the investigator's ability to evaluate the patient's condition or could compromise patient safety. Participation in a clinical trial evaluating an investigational device within 3 months prior to enrollment in this study.
* Stricture length > 5 cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-12-23 (Actual); Primary Completion 2016-09-25 (Actual); Study Completion 2016-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter D. Siersema, MD, Principal Investigator — Study Principal Investigator
Locations (4):
- Instituto do Cancer do Estado de Sao Paulo, São Paulo, Brazil
- Netherlands (2):
  - Erasmus Medical Center, Rotterdam, CE
  - Academisch Medisch Centrum, Amsterdam
- Karolinska Universitets Sjukhuset, Stockholm, Sweden

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metal Stent | Bougie Dilation
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metal Stent | Bougie Dilation | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (6.3) | 66.6 (7.7) | 66.6 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Type of Esophagectomy [Count of Participants; unit: Participants]
  Transthoracic | 6 | 8 | 14
  Transhiatal | 3 | 1 | 4
Maximum Dilation [Mean (Standard Deviation); unit: mm] | 16.4 (0.9) | 15.9 (2.0) | 16.2 (1.5)
Dysphagia Score [Count of Participants; unit: Participants] — Dysphagia Scoring System (scale range from 0 to 4):
  Dysphagia Score = 0: ability to eat a normal diet Dysphagia Score = 1: ability to eat some solids Dysphagia Score = 2: ability to eat some semisolids only Dysphagia Score = 3: ability to swallow liquids only Dysphagia Score = 4: complete dysphagia
  A lower score indicates a better outcome. A higher score indicates a worse outcome.
  Participants
    Dysphagia Score = 2 | 6 | 9 | 15
    Dysphagia Score > 2 | 3 | 0 | 3
Number of Pretreatment Dilations [Mean (Standard Deviation); unit: Pretreatment Dilations] | 2.0 (0.0) | 2.4 (1.0) | 2.2 (0.7)
Quality of Life Overall Health Score [Median (Inter-Quartile Range); unit: units on a scale] — Quality of life scale measuring overall health score. The scale is numbered from 0 to 100. 0 is the worst health the participant can imagine. 100 is the best health the participant can imagine. A lower score indicates a worse outcome. A higher score indicates a better outcome.
  units on a scale | 65.0 [50.0 to 70.0] | 80.0 [70.0 to 80.0] | 70.0 [60 to 80]

OUTCOME MEASURES:

1. Primary Outcome: Number of Dilation Procedures
Description: Number of dilation procedures for the management of dysphagia within 12 months following initial study treatment.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Dilation procedures
Arm/Group | Metal Stent | Bougie Dilation
Number analyzed (Participants) | 9 | 9
Dilation procedures | 5.4 (5.4) | 2.4 (2.5)
Statistical Analysis 1: Comparison: Metal Stent vs Bougie Dilation; Test type: Superiority; p = 0.159, Generalized Linear Model

2. Secondary Outcome: Number of Participants With Technical Stent Placement Success
Description: Technical stent placement success is defined as the ability to deploy the stent in satisfactory position across the stricture.
Time Frame: 12 months
Population: Outcome measure only applicable to participants in the Metal Stent arm, as only participants in the Metal Stent arm received a stent. Participants in the Bougie Dilation arm did not receive a stent and therefore there is no data to collect regarding technical success of stent placement for the Bougie arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Metal Stent | Bougie Dilation
Number analyzed (Participants) | 9 | 0
Participants | 9 | 0

3. Secondary Outcome: Number of Participants With Technical Stent Removal Success
Description: Technical stent removal success is defined as the ability to remove the stent without complications.
Time Frame: 12 months
Population: Outcome measure only applicable to participants in the Metal Stent arm, as only participants in the Metal Stent arm received a stent and therefore underwent stent removal. Participants in the Bougie Dilation arm did not receive a stent and therefore there is no data to collect regarding technical success of stent removal for the Bougie arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Metal Stent | Bougie Dilation
Number analyzed (Participants) | 9 | 0
Participants | 9 | 0

4. Secondary Outcome: Patient's Satisfaction With the Therapy
Description: Patient's satisfaction with the therapy (scored by a visual analog scale) assessed at day 2, week 2, month 1, month 2, month 3, month 6, month 9, and month 12. Patient Satisfaction with Therapy scale ranges from 0-10. The minimum on this scale is 0 (0 being completely unsatisfied with the therapy; a worse outcome) and the maximum on this scale is 10 (10 being completely satisfied with the therapy; a better outcome).
Time Frame: Day 2, Week 2, Month 1, Month 2, Month 3, Month 6, Month 9, and Month 12
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Metal Stent | Bougie Dilation
Number analyzed (Participants) | 9 | 9
score on a scale
  Day 2 | 8.0 [7.0 to 8.0] | 10.0 [8.0 to 10.0]
  Week 2 | 8.0 [8.0 to 9.0] | 9.5 [7.0 to 10.0]
  Month 1 | 9.0 [8.0 to 9.0] | 10.0 [6.0 to 10.0]
  Month 2 | 9.0 [8.0 to 10.0] | 8.0 [8.0 to 10.0]
  Month 3 | 8.0 [8.0 to 9.0] | 8.0 [8.0 to 10.0]
  Month 6 | 8.0 [8.0 to 9.0] | 9.0 [8.0 to 10.0]
  Month 9 | 9.5 [7.5 to 10.0] | 9.0 [7.0 to 10.0]
  Month 12 | 9.0 [7.5 to 10.0] | 10.0 [8.0 to 10.0]

5. Secondary Outcome: Patient's Report of Pain
Description: Patient's report of pain (scored by a visual analog scale) assessed at Baseline, day 2, week 2, month 1, month 2, month 3, month 6, month 9, and month 12. Pain Numerical Rating Scale ranges from 0-10. The minimum on this scale is 0 (0 being no pain; a better outcome) and the maximum on this scale is 10 (10 being worst pain ever; a worse outcome).
Time Frame: Baseline, Day 2, Week 2, Month 1, Month 2, Month 3, Month 6, Month 9, and Month 12
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Metal Stent | Bougie Dilation
Number analyzed (Participants) | 9 | 9
score on a scale
  Baseline | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 2.0]
  Day 2 | 3.0 [1.0 to 4.0] | 0.0 [0.0 to 2.0]
  Week 2 | 1.0 [0.0 to 4.0] | 0.0 [0.0 to 1.0]
  Month 1 | 0.0 [0.0 to 1.0] | 0.0 [0.0 to 1.0]
  Month 2 | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 1.0]
  Month 3 | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 1.0]
  Month 6 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Month 9 | 0.0 [0.0 to 1.5] | 0.0 [0.0 to 0.0]
  Month 12 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

6. Secondary Outcome: Quality Of Life Overall Health Score
Description: Quality of life scale measuring overall health score assessed at day 2, week 2, month 1, month 2, month 3, month 6, month 9, and month 12. The scale is numbered from 0 to 100. 0 is the worst health the participant can imagine. 100 is the best health the participant can imagine. A lower score indicates a worse outcome. A higher score indicates a better outcome.
Time Frame: Day 2, Week 2, Month 1, Month 2, Month 3, Month 6, Month 9, and Month 12
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Metal Stent | Bougie Dilation
Number analyzed (Participants) | 9 | 9
score on a scale
  Day 2 | 70.0 [65.0 to 75.0] | 75.0 [70.0 to 80.0]
  Week 2 | 70.0 [70.0 to 75.0] | 80.0 [60.0 to 80.0]
  Month 1 | 80.0 [75.0 to 85.0] | 80.0 [70.0 to 90.0]
  Month 2 | 80.0 [75.0 to 80.0] | 77.5 [56.0 to 87.5]
  Month 3 | 75.0 [60.0 to 85.0] | 85.0 [70.0 to 90.0]
  Month 6 | 67.5 [62.5 to 75.0] | 85.0 [60.0 to 90.]
  Month 9 | 70.0 [62.5 to 80.0] | 80.0 [70.0 to 90.0]
  Month 12 | 75.0 [67.5 to 85.0] | 70.0 [70.0 to 90.0]

7. Secondary Outcome: Occurrence and Severity of Adverse Events Related to the Stent/Bougie Dilator and/or the Procedure
Description: Occurrence and severity of adverse events related to the stent/bougie dilator and/or the procedure.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metal Stent | Bougie Dilation
Number analyzed (Participants) | 9 | 9
Participants
  Related Serious Adverse Events | 1 | 0
  Related Non-serious Adverse Events | 5 | 0

8. Secondary Outcome: Time to Recurrence of Dysphagia
Description: Time to recurrence of dysphagia, defined as inability of a normal diameter gastroscope (9.8mm) to pass the stricture.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Metal Stent | Bougie Dilation
Number analyzed (Participants) | 9 | 9
Days | 36 [24 to 71] | 33 [21 to 33]

9. Secondary Outcome: Total Number of Stent Migrations
Description: Total number of stent migrations with or without symptoms.
Time Frame: 12 months
Measure: Number; unit: stent migrations
Arm/Group | Metal Stent | Bougie Dilation
Number analyzed (Participants) | 9 | 9
stent migrations | 2 | 0

10. Secondary Outcome: Number of Reinterventions Within 12 Months Following the Initial Study Treatment
Description: Number of reinterventions within 12 months following the initial study treatment.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: reinterventions
Arm/Group | Metal Stent | Bougie Dilation
Number analyzed (Participants) | 9 | 9
reinterventions | 5.6 (5.3) | 2.9 (2.7)

ADVERSE EVENTS:
Time Frame: Adverse event data collected for events related to the stent/bougie dilator and/or the procedure, from the time the participant signed the informed consent and was randomized to the study, until completion of the 12 month follow-up visit (occurring 12 months post-initial study treatment).
Description: Collected and reported only on those Adverse Events (Serious and Non-serious) related to the stent/bougie dilator and/or the procedure.
Arm/Group | Metal Stent | Bougie Dilation
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/9
Other Adverse Events (participants affected / at risk) | 5/9 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metal Stent (N=9) | Bougie Dilation (N=9)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metal Stent (N=9) | Bougie Dilation (N=9)
Recurrent Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Foreign Body Sensation (General disorders) | 1 (1) | 0 (0)
Retching due to Foreign Body Sensation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thoracic Pain (General disorders) | 1 (1) | 0 (0)
Cervical Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days